CLINICAL TRIAL: NCT00005312
Title: International Programs Collaborative Studies Coordinating Center
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4068
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Lung Diseases

SUMMARY:
To continue the work of the Collaborative Studies Coordinating Center (CSCC) on international studies in cardiopulmonary disease epidemiology. The work was being performed under bilateral agreements that the NHLBI had entered into with Russia, The People's Republic of China and Pakistan. The contract provided nutritional, epidemiologic and biostatistical services in support of these studies.

DETAILED DESCRIPTION:
BACKGROUND:

Computer processing, biostatistical, and epidemiological services at the Collaborative Studies Coordinating Center (CSCC) had been funded previously as part of the NHLBI Lipid Research Clinics (LRC) contracts. In FY 1990, contract N01HV08112 was awarded separately from the LRC for the first time and provided services for collaborative studies carried out under NHLBI international bilateral agreements with the USSR, Poland, and the People's Republic of China. The assistance has provided important contributions to large-scale, international epidemiological studies resulting from bilateral agreements between the United States and other countries. The results of these efforts have provided insights into different disease patterns and trends throughout the world.

DESIGN NARRATIVE:

The CSCC coordinated data collection and data file transfer, coordinated scientific meetings, visited the collaborating countries, hosted collaborative scientists, and directed data analysis, combining data from all countries.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-01; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Clarence Davis — University of North Carolina

REFERENCES:
- [Background] Stevens J, Alexandrov AA, Smirnova SG, Deev AD, Gershunskaya YuB, Davis CE, Thomas R. Comparison of attitudes and behaviors related to nutrition, body size, dieting, and hunger in Russian, black-American, and white-American adolescents. Obes Res. 1997 May;5(3):227-36. doi: 10.1002/j.1550-8528.1997.tb00297.x. PMID 9192397
- [Background] Pajak A, Williams OD, Broda G, Baczynska E, Rywik S, Davis CE, Kawalec E, Chodkowska E, Irving S, Manolio T. Changes over time in blood lipids and their correlates in Polish rural and urban populations: the Poland-United States Collaborative Study in cardiopulmonary disease epidemiology. Ann Epidemiol. 1997 Feb;7(2):115-24. doi: 10.1016/s1047-2797(96)00125-1. PMID 9099399
- [Background] Shalnova S, Shestov DB, Ekelund LG, Abernathy JR, Plavinskaya S, Thomas RP, Williams DH, Deev A, Davis CE. Blood pressure and heart rate response during exercise in men and women in the USA and Russia lipid research clinics prevalence study. Atherosclerosis. 1996 Apr 26;122(1):47-57. doi: 10.1016/0021-9150(95)05746-3. PMID 8724111
- [Background] Davis CE, Williams DH, Oganov RG, Tao SC, Rywik SL, Stein Y, Little JA. Sex difference in high density lipoprotein cholesterol in six countries. Am J Epidemiol. 1996 Jun 1;143(11):1100-6. doi: 10.1093/oxfordjournals.aje.a008686. PMID 8633598
- [Background] Broda G, Davis CE, Pajak A, Williams OD, Rywik SL, Baczynska E, Folsom AR, Szklo M. Poland and United States Collaborative Study on Cardiovascular Epidemiology. A comparison of HDL cholesterol and its subfractions in populations covered by the United States Atherosclerosis Risk in Communities Study and the Pol-MONICA Project. Arterioscler Thromb Vasc Biol. 1996 Feb;16(2):339-49. doi: 10.1161/01.atv.16.2.339. PMID 8620351
- [Background] Perova NV, Oganov RG, Williams DH, Irving SH, Abernathy JR, Deev AD, Shestov DB, Zhukovsky GS, Davis CE, Tyroler HA. Association of high-density-lipoprotein cholesterol with mortality and other risk factors for major chronic noncommunicable diseases in samples of US and Russian men. Ann Epidemiol. 1995 May;5(3):179-85. doi: 10.1016/1047-2797(94)00104-2. PMID 7606306
- [Background] Davis CE, Pajak A, Rywik S, Williams DH, Broda G, Pazucha T, Ephross S. Natural menopause and cardiovascular disease risk factors. The Poland and US Collaborative Study on Cardiovascular Disease Epidemiology. Ann Epidemiol. 1994 Nov;4(6):445-8. doi: 10.1016/1047-2797(94)90003-5. PMID 7804498
- [Background] Davis CE, Deev AD, Shestov DB, Perova NV, Plavinskaya SI, Abolafia JM, Kim H, Tyroler HA. Correlates of mortality in Russian and US women. The Lipid Research Clinics Program. Am J Epidemiol. 1994 Feb 15;139(4):369-79. doi: 10.1093/oxfordjournals.aje.a117009. PMID 8109571
- [Background] Dennis BH, Zhukovsky GS, Shestov DB, Davis CE, Deev AD, Kim H, Tyroler HA. The association of education with coronary heart disease mortality in the USSR Lipid Research Clinics Study. Int J Epidemiol. 1993 Jun;22(3):420-7. doi: 10.1093/ije/22.3.420. PMID 8359957
- [Background] Shestov DB, Deev AD, Klimov AN, Davis CE, Tyroler HA. Increased risk of coronary heart disease death in men with low total and low-density lipoprotein cholesterol in the Russian Lipid Research Clinics Prevalence Follow-up Study. Circulation. 1993 Sep;88(3):846-53. doi: 10.1161/01.cir.88.3.846. PMID 8353914
- [Background] Rywik SL, Manolio TA, Pajak A, Piotrowski W, Davis CE, Broda GB, Kawalec E. Association of lipids and lipoprotein level with total mortality and mortality caused by cardiovascular and cancer diseases (Poland and United States collaborative study on cardiovascular epidemiology). Am J Cardiol. 1999 Sep 1;84(5):540-8. doi: 10.1016/s0002-9149(99)00374-4. PMID 10482152
- [Background] Pajak A, Broda G, Manolio TA, Kawalec E, Rywik S, Davis CE, Pikon J, Pytlak A, Thomas RP. Constitutional, biochemical and lifestyle correlates of fibrinogen and factor VII activity in Polish urban and rural populations. Int J Epidemiol. 1998 Dec;27(6):953-61. doi: 10.1093/ije/27.6.953. PMID 10024188
- [Background] Wu Y, Vollmer WM, Buist AS, Tsai R, Cen R, Wu X, Chen P, Li Y, Guo C, Mai J, Davis CE. Relationship between lung function and blood pressure in Chinese men and women of Beijing and Guangzhou. PRC-USA Cardiovascular and Cardiopulmonary Epidemiology Research Group. Int J Epidemiol. 1998 Feb;27(1):49-56. doi: 10.1093/ije/27.1.49. PMID 9563693
- [Background] Rywik SL, Davis CE, Pajak A, Broda G, Folsom AR, Kawalec E, Williams OD. Poland and U.S. collaborative study on cardiovascular epidemiology hypertension in the community: prevalence, awareness, treatment, and control of hypertension in the Pol-MONICA Project and the U.S. Atherosclerosis Risk in Communities Study. Ann Epidemiol. 1998 Jan;8(1):3-13. doi: 10.1016/s1047-2797(97)00177-4. PMID 9465988
- [Background] Perova NV, Davis CE, Tao S, Pajak A, Stein Y, Broda GB, Li Y, Tyroler HA. Multi-country comparison of plasma lipid relationship to years of schooling in men and women. Int J Epidemiol. 2001 Apr;30(2):371-9. doi: 10.1093/ije/30.2.371. PMID 11369745
- [Background] Rywik SL, Williams OD, Pajak A, Broda G, Davis CE, Kawalec E, Manolio TA, Piotrowski W, Hutchinson R. Incidence and correlates of hypertension in the Atherosclerosis Risk in Communities (ARIC) study and the Monitoring Trends and Determinants of Cardiovascular Disease (POL-MONICA) project. J Hypertens. 2000 Aug;18(8):999-1006. doi: 10.1097/00004872-200018080-00002. PMID 10953989
- [Background] Dennis BH, Pajak A, Pardo B, Davis CE, Williams OD, Piotrowski W. Weight gain and its correlates in Poland between 1983 and 1993. Int J Obes Relat Metab Disord. 2000 Nov;24(11):1507-13. doi: 10.1038/sj.ijo.0801435. PMID 11126349
- [Background] Burke GL, Rywik S, Pajak A, et al: Mortality attributable to hypertension in Eastern Europe compared to the United States. CVD Prevention, 3:213-220, 2000.
- [Background] Li YH, Li Y, Davis CE, Chen Z, Tao S, Folsom AR, Bachorik P, Stamler J, Abernathy JR. Serum cholesterol changes from 1983-1984 to 1993-1994 in the People's Republic of China. Nutr Metab Cardiovasc Dis. 2002 Jun;12(3):118-26. PMID 12325468